CLINICAL TRIAL: NCT00083785
Title: Safety and Effectiveness of Treating Cancers With the Litx™ System and Chemotherapy. Section A: Phase II Safety and Effectiveness Study in Patients With Liver Metastases From Colorectal Cancer
Brief Title: Study of the Litx™ System Combined With Chemotherapy in Patients With Colorectal Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSC-OL003
Record Dates: First submitted 2004-06-02; First posted 2004-06-03 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Liver Metastasis; Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis | interventions — Talaporfin; Photochemotherapy; Phototherapy; Drug Therapy

INTERVENTIONS:
Drug: Talaporfin sodium (LS11)
Device: LED-based light infusion device
Device: Light emitting diodes (LED)
Procedure: Photodynamic therapy
Procedure: Phototherapy
Procedure: Chemotherapy

SUMMARY:
The purpose of this study is to determine whether the Litx™ system is safe and effective in combination with chemotherapy in the treatment of liver metastasis arising from colorectal cancer. Litx™ is a next-generation photodynamic therapy platform in which the drug, talaporfin sodium (LS11), is activated by light from the light-emitting diode (LED)-based light infusion device, inserted directly into the tumor through the skin prior to treatment.

DETAILED DESCRIPTION:
Patients that provide Informed Consent and satisfy the Eligibility Criteria will undergo CT or Ultrasound guided percutaneous placement of a single, two, three, or four Light Sources depending on their tumor characteristics. No more than 4 Light Sources will be used at a single treatment. The Light Sources may be used in a single lesion or in multiple lesions.

Following radiographic confirmation of Light Source placement, patients will receive an intravenous dose of LS11 at 40 mg/m². Fifteen minutes to 1 hour following completion of LS11 administration, delivery of 200 J/cm at 20 mW/cm light energy will begin. The Light Source will then be manually removed and the patients will be observed for acute complication of Light Source removal. Precautions for protection from external light exposure should be instituted beginning with the LS11 administration and be maintained as defined throughout the study period. On day 3 following Litx™ treatment the patient will receive a standard chemotherapy with Irinotecan or Oxaliplatin with or without 5FU and /or leucovorin for metastatic colorectal cancer. On day 30+5 and day 60+5 the patient will undergo clinical assessment and the tumor mass will be imaged using contrast enhanced spiral CT for determination of volume and radius of PDT necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic liver lesions from colorectal disease
* Biopsy proven evidence of colorectal cancer
* Patients with 4 or fewer lesions greater than 1 cm and with no single lesion greater than 7 cm in maximum diameter
* Age greater than or equal to 18 years
* Patients must be able to sign informed consent
* Life expectancy greater than or equal to 3 months
* ECOG performance status 0-2
* Patients with extrahepatic disease in addition to their hepatic metastases may be eligible
* Must have recovered from the toxicity from any prior antineoplastic therapy

Exclusion Criteria:

* Patients who are candidates for complete surgical resection
* Pregnancy or breast-feeding. A negative pregnancy test (urine or serum) is required prior to enrollment
* Known uncontrollable serious reactions such as anaphylaxis, to the contrast agents used in this study
* PT or PTT greater than 1.5X control
* Platelet count less than 100,000
* WBC less than 2500/mm
* Neutrophils less than 2000/mm
* Hemoglobin less than 9 g/dL
* Liver enzymes (AST, ALT, GGT, alkaline phosphatase) greater than 3 X ULN
* Total bilirubin greater than 1.5 X ULN
* Serum creatinine greater than 2.5 X ULN
* Patients who have been treated with either AVASTIN™ (Bevacizumab) or ERBITUX™ (Cetuximab) within the previous 4 weeks (28 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Lustig RA, Vogl TJ, Fromm D, Cuenca R, Alex Hsi R, D'Cruz AK, Krajina Z, Turic M, Singhal A, Chen JC. A multicenter Phase I safety study of intratumoral photoactivation of talaporfin sodium in patients with refractory solid tumors. Cancer. 2003 Oct 15;98(8):1767-71. doi: 10.1002/cncr.11708. PMID 14534895
- [Background] Chen J, Keltner L, Christophersen J, Zheng F, Krouse M, Singhal A, Wang SS. New technology for deep light distribution in tissue for phototherapy. Cancer J. 2002 Mar-Apr;8(2):154-63. doi: 10.1097/00130404-200203000-00009. PMID 11999949
- See also: Sponsor website — http://www.lightsciences.com